CLINICAL TRIAL: NCT01311245
Title: Testing Stage Tailored vs. Non-stage Tailored Interventions Among Job-seekers With Risky Drinking
Brief Title: Testing Alcohol Interventions Among Job-seekers
Acronym: TOPAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Dr. Jennis Freyer-Adam, Principle Investigator, University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DM5-IESO03; FR2661/1-1 (Other Grant/Funding Number: German Research Foundation); FR2661/1-2 (Other Grant/Funding Number: German Research Foundation); DM5-IESO05 (Registry Identifier: University Medicine Greifswald)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hazardous Drinking
Keywords: Risky drinking; Brief intervention; Computer-generated feedback; Stage-tailored; Non-stage-tailored

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stage-tailored (Experimental): At baseline and three months later
  Interventions: Behavioral: Stage-tailored intervention
- Non-stage-tailored (Experimental): At baseline and three months later
  Interventions: Behavioral: Non-stage-tailored Intervention
- Control group (No Intervention): Assessment only

INTERVENTIONS:
Behavioral: Stage-tailored intervention — Based on the Trans-Theoretical Model of intentional behavior change (TTM). According to their stage of change, participants received two computer generated feedback letters on their risky drinking, stage of change, processes of change, self-efficacy, and decisional balance. The first letter included normative feedback (interpersonal comparison with other individuals in the same stage), and was sent out by mail after baseline. The second letter included normative and ipsative feedback (intrapersonal comparisons: baseline vs. 3 months later), and was sent out by mail three months later.
  Arms: Stage-tailored
Behavioral: Non-stage-tailored Intervention — Based on the Theory of Planned Behavior (TPB). Participants received two computer generated feedback letters on their risky drinking, beliefs (behavioral, normative, control), attitude, subjective norm, perceived behavioral control, intention, and they were asked to fill in a where-when-how to change plan. The first letter included normative feedback (interpersonal comparison with other women/ men), and was sent out by mail after baseline. The second letter included normative and ipsative feedback, and was sent out by mail three months later.
  Arms: Non-stage-tailored

SUMMARY:
The aim of the randomized controlled trial was to test two behavioral interventions among job-seekers with risky drinking. The interventions differed in their theoretical background: Intervention A was tailored to the stage of change, and Intervention B was non-stage-tailored. Over 12 months, job-seekers were pro-actively screened for risky drinking at three job-agencies. Job-seekers with risky drinking were asked to participate in the study. All three groups were assessed at baseline, and 3, 6 and 15 months later. The baseline assessment was self-administered using handheld computers. The follow-up assessments by interviews on the phone, primarily. Both intervention groups received individualized computer generated feedback letters at baseline and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Job-seekers with risky drinking (AUDIT-C ≥ 4/5 [women/men] and AUDIT < 20)

Exclusion Criteria:

* Job-seekers already asked to participate during an earlier visit at the job agency
* Job-seekers not intending to talk to a job-agent/ without waiting time
* Job-seekers physically or mentally not capable of participating in the study
* Job-seekers with insufficient language/ reading skills
* Job-seekers with more severe alcohol problems (AUDIT ≥ 20)
* Job-seekers employed at the department conducting the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1243 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Risky drinking | 6 and 15 months
  Determined by using average alcohol consumption per day, heavy occasional drinking, the Alcohol Use Disorder Identification Test-Consumtion (AUDIT-C) score

SECONDARY OUTCOMES:
Motivation to reduce drinking | 6 and 15 months
  Assessed by the Readiness to Change Questionnaire
Attempts to reduce drinking | 6 and 15 months
Knowledge about drinking limits | 6 and 15 months
Alcohol related problems | 6 and 15 months
Self-rated health | 6 and months

CONTACTS AND LOCATIONS:
Overall Officials: Jennis Freyer-Adam, PhD, Principal Investigator — Institute of Social Medicine and Prevention, University Medicine Greifswald
Locations (3):
- Germany (3):
  - Agentur für Arbeit, Greifswald
  - Agentur für Arbeit, Stralsund
  - Arbeitsgemeinschaft, Stralsund

REFERENCES:
- [Result] Freyer-Adam J, Gaertner B, Tobschall S, John U. Health risk factors and self-rated health among job-seekers. BMC Public Health. 2011 Aug 19;11:659. doi: 10.1186/1471-2458-11-659. PMID 21854611
- [Result] Baumann S, Gaertner B, Schnuerer I, Bischof G, John U, Freyer-Adam J. How well do TTM measures work among a sample of individuals with unhealthy alcohol use that is characterized by low readiness to change? Psychol Addict Behav. 2013 Sep;27(3):573-83. doi: 10.1037/a0029368. Epub 2012 Aug 6. PMID 22867296
- [Result] Freyer-Adam J, Baumann S, Schnuerer I, Haberecht K, Bischof G, John U, Gaertner B. Does stage tailoring matter in brief alcohol interventions for job-seekers? A randomized controlled trial. Addiction. 2014 Nov;109(11):1845-56. doi: 10.1111/add.12677. Epub 2014 Aug 1. PMID 24981701
- [Result] Haberecht K, Schnuerer I, Gaertner B, John U, Freyer-Adam J. The Stability of Social Desirability: A Latent Change Analysis. J Pers. 2015 Aug;83(4):404-12. doi: 10.1111/jopy.12112. Epub 2014 Aug 19. PMID 25041464
- [Result] Baumann S, Gaertner B, Schnuerer I, Haberecht K, John U, Freyer-Adam J. The impact of a stage tailored intervention on alcohol use trajectories among those who do not intend to change. Drug Alcohol Depend. 2015 Feb 1;147:167-74. doi: 10.1016/j.drugalcdep.2014.11.020. Epub 2014 Dec 3. PMID 25500129
- [Result] Schnuerer I, Baumann S, Haberecht K, Gaertner B, John U, Freyer-Adam J. Patterns of health risk behaviors among job-seekers: a latent class analysis. Int J Public Health. 2015 Jan;60(1):111-9. doi: 10.1007/s00038-014-0623-1. Epub 2014 Dec 23. PMID 25532553
- [Result] Baumann S, Gaertner B, Schnuerer I, Haberecht K, John U, Freyer-Adam J. Belief incongruence and the intention-behavior gap in persons with at-risk alcohol use. Addict Behav. 2015 Sep;48:5-11. doi: 10.1016/j.addbeh.2015.04.007. Epub 2015 Apr 18. PMID 25930010
- See also: German Research Foundation — http://www.dfg.de/en/index.jsp